CLINICAL TRIAL: NCT00065897
Title: Randomized Trial of 11-14 Week Amniocentesis and Transabdominal Chorionic Villus Sampling (TA CVS)
Brief Title: Prenatal Testing: Amniocentesis Versus Transabdominal Chorionic Villus Sampling (TA CVS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 5R01HD031991 (NIH); 1R01HD032109 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: Pregnancy
Keywords: Amniocentesis; Transabdominal chorionic villus sampling; Fluorescence in situ hybridization; Alpha fetoprotein; Acetylcholinesterase; Prenatal testing; Prenatal diagnosis
MeSH Terms: conditions — Pain | interventions — Amniocentesis

INTERVENTIONS:
Procedure: Amniocentesis
Procedure: Transabdominal chorionic villus sampling (TA CVS)

SUMMARY:
Prenatal diagnosis can provide information to parents about specific fetal disorders. However, invasive prenatal diagnostic procedures are associated with risks to the fetus. This study will compare the safety and effectiveness of two methods of invasive prenatal diagnosis: amniocentesis and transabdominal chorionic villus sampling (TA CVS).

DETAILED DESCRIPTION:
Amniocentesis is generally performed at 105 to 125 days post last menstrual period (LMP) and TA CVS at 63 to 76 days post LMP. This study will compare the safety and accuracy of transabdominal amniocentesis and TA CVS, each performed during the same modified gestational age window of 77 to 104 days post LMP.

Healthy, pregnant women at 77 to 104 days gestation, whose only indication for prenatal diagnosis is advanced maternal age of at least 34 years at enrollment, will be randomized to receive either TA CVS or amniocentesis following a baseline ultrasound. Eligible women who refuse randomization or for whom a procedure cannot be scheduled by 104 days will also be followed. Primary outcomes include fetal loss or preterm delivery before 196 days gestation as well as total fetal loss, amniotic fluid loss, gestational age at delivery, perinatal morbidity, neonatal morbidity, and congenital abnormalities, including limb reduction defects. Success in obtaining a diagnosis from the two procedures will be compared. One ancillary study will evaluate the feasibility and accuracy of fluorescence in situ hybridization (FISH) as a rapid diagnostic method for certain cytogenetic abnormalities; another will collect data on amniotic fluid alphafetoprotein and acetylcholinesterase for the diagnosis of neural tube defects.

ELIGIBILITY:
Inclusion Criteria

* Singleton pregnancy confirmed by baseline ultrasound
* At least 77 days gestation but not more than 104 days gestation confirmed by baseline ultrasound

Exclusion Criteria

* Evidence of "vanishing" twin
* Bleeding equivalent to a menstrual period at any time during this pregnancy
* Medical history indicating serious maternal illness or potential teratogenic exposure
* Oligohydramnios
* Known fetal abnormality
* Dating inconsistency: if the estimated gestation is 8 or more days less than estimated by LMP, the patient is excluded unless interval growth by ultrasound confirms the normalcy of the pregnancy

Ages: 34 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6400
Dates: Start 1996-09; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Overall Officials: Laird G. Jackson, M.D., Principal Investigator — Drexel University College of Medicine

REFERENCES:
- [Background] Jackson LG, Zachary JM, Fowler SE, Desnick RJ, Golbus MS, Ledbetter DH, Mahoney MJ, Pergament E, Simpson JL, Black S, et al. A randomized comparison of transcervical and transabdominal chorionic-villus sampling. The U.S. National Institute of Child Health and Human Development Chorionic-Villus Sampling and Amniocentesis Study Group. N Engl J Med. 1992 Aug 27;327(9):594-8. doi: 10.1056/NEJM199208273270903. PMID 1640952
- [Background] Elejalde BR, de Elejalde MM, Acuna JM, Thelen D, Trujillo C, Karrmann M. Prospective study of amniocentesis performed between weeks 9 and 16 of gestation: its feasibility, risks, complications and use in early genetic prenatal diagnosis. Am J Med Genet. 1990 Feb;35(2):188-96. doi: 10.1002/ajmg.1320350210. PMID 2309757